CLINICAL TRIAL: NCT02350335
Title: Transdermal Nicotine Replacement in Smokers With Acute Aneurysmal Subarachnoid Hemorrhage
Acronym: NRT-SAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Angelika Sorteberg, Md, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-2561b
Record Dates: First submitted 2015-01-12; First posted 2015-01-29 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: aneurysm; nicotine replacement therapy; cerebral vasospasm; outcome
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm; Vasospasm, Intracranial | interventions — Nicotine; Administration, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NRT (Active Comparator): Active smokers with acute aneurysmal hemorrhage randomly assigned to transdermal nicotine replacement after securing of the aneurysm.
  Patient management for all patients is according to the institutional treatment guidelines and independent of group assignment.
  The dose is dependent on smoke consumption prior to the ictus. Nicorette 7 mg/day for smokers smoking 1-10 cigarettes /day Nicorette 14mg/day for smokers smoking 11-19 cigarettes/day Nicorette 21 mg/day for smokers smoking 20 or more cigarettes daily
  Interventions: Drug: Nicotine (transdermal)
- no NRT (No Intervention): Active smokers with acute aneurysmal hemorrhage that were assigned to not receive transdermal nicotine replacement.
- non-smokers (No Intervention): Non-smokers with acute aneurysmal hemorrhage. Non-smokers do not receive transdermal nicotine replacement. This group is to be compared to the group of active smokers receiving transdermal nicotine replacement and to the group of active smokers not receiving transdermal nicotine replacement.

INTERVENTIONS:
Drug: Nicotine (transdermal) — Application of transdermal nicotine replacement in smokers with acute aneurysmal hemorrhage
  Other Names: Nicotinelle
  Arms: NRT

SUMMARY:
All patients with acute aneurysmal hemorrhage are treated in accordance with our institutional protocol. After securing of the aneurysm, some smokers with acute aneurysmal hemorrhage are randomly assigned to transdermal nicotine replacement (NRT). The short- and long-term effect of NRT will be studied comparing non-smokers, smokers without NRT and smokers with NRT.

DETAILED DESCRIPTION:
Various aspects of the study:

* Study cerebral circulation with transcranial Doppler ultrasonography (TCD) prior to and after NRT.
* Study cardiac output and peripheral vessel resistance minimally invasive (LiDCO) prior to and after NRT in patients that already have established LiDCO.
* Monitor intracranial pressure prior to and after NRT in patients that have established an intracranial pressure sensor.
* Register the frequency of cerebral vasospasm and complications in non-smokers, smokers without NRT, and smokers with NRT.
* Register the use of opioids, opioidanesthetics, propofol og psycholeptics in non-smokers, smokers without NRT, and smokers with NRT.

ELIGIBILITY:
Inclusion Criteria:

* aneurysmal subarachnoid hemorrhage after securing of the aneurysm and surviving the first 2 weeks.

Exclusion Criteria:

* manifest cerebral vasospasm at arrival at our department (i.e. before securing of the aneurysm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cerebral vasospasm | 21 days
  Frequency of cerebral vasospasm within 21 days after the ictus. The institutional protocol for management of aneurysmal hemorrhage is followed in diagnosing cerebral vasospasm. This includes monitoring for cerebral vasospasm with transcranial Doppler ultrasonography and a cerebral computed tomography angiogram on day 7 after the ictus. Digital subtraction angiography is performed when necessary. All patients are monitored in the intensive care or intermediate care unit for clinical signs of cerebral vasospasm.

SECONDARY OUTCOMES:
Smoking status | 1 year
  Managed to quit smoking after NRT?
Functional outcome | 3 and 12 months
  Glasgow outcome scale, Glasgow outcome scale extended, Rankin Stroke Scale, return to work
Drug consumption | as long as the patient is in the intensive care unit
  Use of sedatives and anesthetics
Cerebral infarction | 3-6 months
  Radiological evidence of irreversible brain tissue damage. All patients have a control scan approximately 3 months after the ictus. This is either a computed tomography scan (if the patient had the aneurysm secured surgically) or a magnetic resonance image (if the patient had endovascular repair of the aneurysm)
Complications | 3-6 months
  Frequency of complications including secondary hydrocephalus and mortality. Special emphasis on thrombo-embolic complications (deep venous thrombosis and pulmonary embolism)

CONTACTS AND LOCATIONS:
Overall Officials: Angelika G Sorteberg, MD, PhD, Principal Investigator — Consulting neurosurgeon, Head of division Rikshospitalet
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seder DB, Schmidt JM, Badjatia N, Fernandez L, Rincon F, Claassen J, Gordon E, Carrera E, Kurtz P, Lee K, Connolly ES, Mayer SA. Transdermal nicotine replacement therapy in cigarette smokers with acute subarachnoid hemorrhage. Neurocrit Care. 2011 Feb;14(1):77-83. doi: 10.1007/s12028-010-9456-9. PMID 20949331
- [Background] Krishnamurthy S, Kelleher JP, Lehman EB, Cockroft KM. Effects of tobacco dose and length of exposure on delayed neurological deterioration and overall clinical outcome after aneurysmal subarachnoid hemorrhage. Neurosurgery. 2007 Sep;61(3):475-80; discussion 480-1. doi: 10.1227/01.NEU.0000290892.46954.12. PMID 17881958
- [Background] Weir BK, Kongable GL, Kassell NF, Schultz JR, Truskowski LL, Sigrest A. Cigarette smoking as a cause of aneurysmal subarachnoid hemorrhage and risk for vasospasm: a report of the Cooperative Aneurysm Study. J Neurosurg. 1998 Sep;89(3):405-11. doi: 10.3171/jns.1998.89.3.0405. PMID 9724114